CLINICAL TRIAL: NCT04835766
Title: Urodynamic Changes Following Bladder Injury During Surgical Management of Placenta Accreta Spectrum: A Multicenter Study
Brief Title: Urodynamic Changes Following Bladder Injury
Acronym: Uro-PAS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ayman S Dawood, MD, Assistant professor, Tanta University
Other Study IDs: Uro-PAS
Record Dates: First submitted 2021-04-02; First posted 2021-04-08 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Urologic Injuries; Urodynamic Changes; Bladder Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Symptomatic group: These patients had bladder injury during PAS surgery and had Lower urinary tract symptoms
  Interventions: Diagnostic Test: Urodynamic study
- Asymptomatic group: These patients had bladder injury during PAS surgery and had no Lower urinary tract symptoms
  Interventions: Diagnostic Test: Urodynamic study

INTERVENTIONS:
Diagnostic Test: Urodynamic study — Uroflowmetry, voiding cystometrogram, maximum flow rate (Qmax) and detrusor pressure at maximum flow (Pdet Qmax).

SUMMARY:
This study is a unique one as it si done for first time to all patients following bladder injury in PAS surgery. Bladder function will be assessed by urodynamic study.

DETAILED DESCRIPTION:
Patients will be initially assessed by overactive bladder (OAB) and incontinence questionnaire. Examination was done to determine any neurological, or congenital abnormalities.

Urodynamic study (UDS) will done for all patients. The patients will be asked to drink fluids to obtain a comfortably full bladder. Initially, a pelvic-abdominal ultrasound was done followed by the UDS. Urodynamic study consisted of uroflowmetry (volume: ≥150 ml and Qmax: 20-30 ml/s); filling cystometry in physiological or medium filling rate of 40 ml/min (using normal saline at room temperature through a double lumen urethral catheter); stress leak test; and pressure flow study.

No sedation will be administered during the study as the patient should be aware. The patients were placed in a semi-seated lithotomy position. After a detailed explanation to the patient, the examination will begin by passing a catheter into the bladder (5 Fr) to measure the postvoiding residual urine followed by filling the bladder and measuring the intravesical pressure through the catheter.

A rectal catheter was placed for measuring the abdominal pressure. The systems will be always zeroed at the atmospheric pressure. The patients will be periodically asked to cough to check the operation of the equipment and instructed to report her sensations.

The volume of the first sensation of filling, first desire (1 s) and second desire (2 s) were recorded. When the bladder was filled up to 150 ml, patients were asked to cough (Valsalva) to predict the stress leakage. If not occur at 150 ml, the bladder was refilled, and the stress test was repeated until the leakage occurred or the bladder capacity was reached. Additionally, any unidentified involuntary detrusor contractions will be noted.

When the patient had the urge to void, the permission for voiding will be given. Then voiding cystometrogram (pressure-flow) was performed and the urodynamic parameters, such as maximum flow rate (Qmax) and detrusor pressure at maximum flow (Pdet Qmax) will be observed.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-40 years
* Placenta accreta managed either by cesarean hysterectomy or by uterine sparing conservative treatment
* Bladder injury was diagnosed and repaired during surgery 6 months ago.

Exclusion Criteria:

* Patients with neurological problems
* Presence of congenital urinary system anomalies
* Urinary tract infections (UTIs)
* Previous urologic surgeries
* Patients with stone bladder or tumour
* Diabetic patients

Ages: 20 Years to 40 Years | Sex: Female
Age Groups: Adult
Study Population: This study is multi-center descriptive cohort study. This study will be conducted at Urology departments. Cases were recruited from both Obstetrics and gynecology and Urology departments of Al-Azhar University and Tanta University. All cases had past history of bladder injury during PAS surgery either by hysterectomy or uterine sparing techniques.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Bladder dysfunction | 6 months
  Uroflowmerty measuring the flow of urine in ml per minute
Residual urine volume | 6 months
  Assessed by ultrasound to measure volume of residual urine
maximum flow rate | 6 months
  Urodynamic study
Detrusor pressure at maximum flow | 6 months
  Urodynamic study

CONTACTS AND LOCATIONS:
Locations (1):
- Ayman Shehata Dawood, Tanta, Algharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
On request
Supporting Information: Study Protocol
Time Frame: 3 months